CLINICAL TRIAL: NCT00674284
Title: Change of Serum Cortisol Levels in Patients Without Improvement in Intensive Care Unit
Brief Title: Adrenal Exhaustion Syndrome in Critically Ill Patients Without Improvement
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chao-Chi Ho, National Taiwan University Hospital
Other Study IDs: 200802022R
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We study the relationship between patient outcomes and sequential changes of serum cortisol level.

DETAILED DESCRIPTION:
Elevated corticosteroid level to meet physiologic needs during acute illness is a protective response for stress. This homeostasis is maintained by the hypothalamic-pituitary-adrenal (HPA) axis. However, inadequate response as corticosteroid insufficiency in critically ill patients is reported with increasing frequency, especially in severe sepsis and septic shock. Thus, corticosteroids could be beneficial for septic shock or severe acute illness.

Once considered as normal adrenal function, adrenal insufficiency may developed later with chronic critical illness as adrenal exhaustion syndrome. It is easily overlooked and is possible due to the chronic secretion of systemic cytokines or other HPA axis-suppressive substances. There is still no consensus how often adrenal function testing should be repeated, although a re-evaluation should be considered if clinical symptoms and signs suggest adrenal insufficiency or deteriorating clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* ICU admission
* had two cortisol data

Exclusion Criteria:

* first cortisol data abnormal
* cortisol data not checked in ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of the adult patients (age >18 years) admitted to the intensive care units of the National Taiwan University Hospital between January 2005 and December 2006 were surveyed.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, MD, Study Director — 1. Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Chao-Chi Ho, Taipei, Taiwan